CLINICAL TRIAL: NCT01364155
Title: A Randomized, Single-Blind, Placebo-Controlled Phase 2 Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LIM-0705 in Subjects With Impaired Glucose Tolerance or Abnormal HOMA-IR
Brief Title: Safety, Tolerability, PK, and PD of LIM-0705 in Subjects With Impaired Glucose Tolerance or Abnormal HOMA-IR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Limerick BioPharma (Industry)
Responsible Party: Linda Morrow, MD, Profil Institute for Clinical Research, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIM-0705-CL-2001
Record Dates: First submitted 2011-05-25; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Impaired Glucose Tolerance; Insulin Resistance
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 600 mg LIM-0705 BID for 28 days (Experimental)
  Interventions: Drug: LIM-0705
- Placebo LIM-0705 for 28 days (Placebo Comparator)
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: LIM-0705
  Arms: 600 mg LIM-0705 BID for 28 days
Drug: Placebo capsules
  Arms: Placebo LIM-0705 for 28 days

SUMMARY:
Preliminary research suggests that LIM-0705 improves insulin sensitivity with neutral effects on weight in obese and diabetic rodent models. Results from a Phase 1b clinical study, conducted in healthy volunteers, indicate that LIM-0705 and a major metabolite may be potential insulin sensitizers by OGTT.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety and tolerability of LIM-0705 administered for 28 days in adult males and females with impaired glucose tolerance or abnormal HOMA-IR.

Secondary Objectives include:

* examine the pharmacokinetics (PK) of LIM-0705
* explore the pharmacodynamics (PD) of LIM-0705 in obese adult males and females with impaired glucose tolerance (defined as two-hour plasma glucose levels of ≥140 to ≤199 mg per dL [7.8 to 11.06 mmol/L] on the 75-g oral glucose tolerance test [OGTT]) or abnormal HOMA-IR (HOMA-IR value ≥ 2.5) as measured by change in response to hyperinsulinemic clamp, mixed-meal tolerance test (MMTT) between Days -2 and 27
* explore the effect of LIM-0705 on fasting lipid, insulin and glucose profiles compared to baseline levels

ELIGIBILITY:
Inclusion Criteria:

* males and females, age 18-75 years old, able and willing to provide written informed consent to participate in the study
* obesity-induced impaired glucose tolerance or abnormal HOMA-IR
* waist circumference of 40 inches or greater (men) or 35 inches or greater (women)
* good physical health based on EKG, electrolytes, LDH, creatinine, urea, AST, ALT, alkaline phosphatase, and renal function
* male subjects who are sexually active with a female partner of childbearing age must agree to use of 2 effective methods of contraception, including the use of a condom, throughout the course of the study or provide proof of surgical sterility. The second method of contraception must be the use by their female partners of any of the following: a diaphragm with spermicide, a cervical cap with spermicide, an IUD, a female condom, or an approved hormonally based contraceptive (e.g., an oral, transdermal, or implanted estrogen or progestin). Female subjects must be post menopausal or surgically sterile.

Exclusion Criteria:

* BMI equal to or greater than 40 kg/m2
* allergy to onions or red wine
* strict vegetarians
* use of any non-study medications other than thyroid replacement hormone or anti-hypertensives. Use of cardesarten cilexetil is not permitted. Note: acetaminophen should not be administered.
* use of chemotherapy agents or history of cancer, other than non-metastatic non-melanoma skin cancer that has been completely excised, within 5 years prior to the screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety (number of subjects with adverse events) of LIM-0705 administered to adult males and females with impaired glucose tolerance or abnormal HOMA-IR | 28 days

SECONDARY OUTCOMES:
Examine the pharmacokinetics (PK) of LIM-0705 as measured by area under the curve (AUC). | 28 days
Explore the pharmacodynamics (PD) of LIM-0705 in obese adult males and females with impaired glucose tolerance or abnormal HOMA-IR as measured by change in response to hyperinsulinemic clamp, mixed-meal tolerance test (MMTT) between Days -2 and 27 | 28 days
Explore the effect of LIM-0705 on fasting lipid, insulin and glucose profiles compared to baseline levels | 28 days
Evaluate the tolerability (BID) of LIM-0705 administered to adult males and females with impaired glucose tolerance or abnormal HOMA-IR | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Linda Morrow, MD, Principal Investigator — Profil Institute of Clinical Research, Inc.
Locations (1):
- Profil Institute of Clinical Research, Inc., Chula Vista, California, United States